CLINICAL TRIAL: NCT05791357
Title: The Role of Polymerase Chain Reaction in the Management of Patients With Infective Endocarditis: Modern Diagnostic and Therapeutic Concepts
Brief Title: The Role of Polymerase Chain Reaction in the Management of Patients With Infective Endocarditis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3451
Record Dates: First submitted 2023-02-27; First posted 2023-03-30 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-02

CONDITIONS: Endocarditis Infective
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endocarditis patients (Experimental): Patients with endocarditis who respect including criteria
  Interventions: Diagnostic Test: PCR (Polymerase Chain Reaction) targeting the 16 ribosomal DNA

INTERVENTIONS:
Diagnostic Test: PCR (Polymerase Chain Reaction) targeting the 16 ribosomal DNA — Molecular diagnostic using a broad range PCR on obtained histological material (native valve/valve prosthesis/fragments of them)

SUMMARY:
The aim of this study is to prospectively investigate the additional diagnostic value of broad range PCR targeting the 16 ribosomal DNA in diagnosis and management of patients with infective endocarditis who are candidate for surgicaltherapy;

DETAILED DESCRIPTION:
Study protocol is divided into four different phases:screening, pre-operative clinical assessment (T-1), cardiac surgery (T0) and follow-up period (T4 eT90).

During the screening phase, patients will be assessed to determine whether they met the study inclusion/exclusion criteria. After signing the informed consent, patients will go through a preoperative clinical evaluation (T-1). The following assessments are carried out the day before surgery: recording patient's generality, present antibiotic therapy and possible results of blood cultures performed prior to recruitment; - Twelve-lead ECG; - chest X-ray - transthoracic echocardiogram (TTE); -. three pairs of blood cultures from three different blood sampling sites. In cases of complicated endocarditis, the presence and location of septic embolisms is recorded (using Total body CT scan imaging), signs of heart failure evaluated and operability criteria are assessed. On the day of cardiac surgery (T0), main intraoperative data (valve findings, type of prosthesis, surgery time, cardiopulmonary bypass time and aortic cross clamping time) will be gathered; the excised valve was sent partly to the microbiology laboratory for culture and molecular tests and partly to the pathology Laboratory.

After cardiac surgery, patients continued to be monitored for a follow up at four (T4) and 90 (T90) days after surgery. During the follow-up period, information was collected on the patient's clinical status (vital parameters) and the antibiotic treatment performed. The same blood tests performed at T-1 are repeated at T4 and T90. All this data was recorded on a dedicated database.

ELIGIBILITY:
Inclusion Criteria:

1. patients older than 18 years, with diagnosis of IE on a native or prosthetic valve and with a surgical indication for heart valve replacement using extracorporeal circulation (CPB).
2. patients who have signed informed consent to the partecipation of the study

Exclusion criteria:

1. patients younger than 18 years
2. Failure to sign consent for personal data processing and/or study participation
3. Participation in other experimental studies
4. Patients who did not complete the examinations under study (culture test on blood and excised valve, molecular tests)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Impact of molecular diagnostic tests on the identification of microorganisms | through study completion, an average of 1 year
  number of patients with positive blood cultures vs number of patients with negative blood cultures but with positive molecular diagnostic tests
number of microorganism isolated | through study completion, an average of 1 year
  number of microorganism isolated through molecular diagnostic tests

SECONDARY OUTCOMES:
Impact of molecular diagnostic tests on antibiotic therapy | through study completion, an average of 1 year
  Number of patients with IE in which antibiotic therapy change because of the results of molecular diagnostic tests

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Massetti, Principal Investigator — Fondazione Universitaria Policliino Gemelli IRCSS
Locations (2):
- Italy (2):
  - IRCCS Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Policlinico Agostino Gemelli, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cahill TJ, Baddour LM, Habib G, Hoen B, Salaun E, Pettersson GB, Schafers HJ, Prendergast BD. Challenges in Infective Endocarditis. J Am Coll Cardiol. 2017 Jan 24;69(3):325-344. doi: 10.1016/j.jacc.2016.10.066. PMID 28104075
- [Background] Habib G, Lancellotti P, Antunes MJ, Bongiorni MG, Casalta JP, Del Zotti F, Dulgheru R, El Khoury G, Erba PA, Iung B, Miro JM, Mulder BJ, Plonska-Gosciniak E, Price S, Roos-Hesselink J, Snygg-Martin U, Thuny F, Tornos Mas P, Vilacosta I, Zamorano JL; ESC Scientific Document Group. 2015 ESC Guidelines for the management of infective endocarditis: The Task Force for the Management of Infective Endocarditis of the European Society of Cardiology (ESC). Endorsed by: European Association for Cardio-Thoracic Surgery (EACTS), the European Association of Nuclear Medicine (EANM). Eur Heart J. 2015 Nov 21;36(44):3075-3128. doi: 10.1093/eurheartj/ehv319. Epub 2015 Aug 29. No abstract available. PMID 26320109
- [Background] Baddour LM, Wilson WR, Bayer AS, Fowler VG Jr, Tleyjeh IM, Rybak MJ, Barsic B, Lockhart PB, Gewitz MH, Levison ME, Bolger AF, Steckelberg JM, Baltimore RS, Fink AM, O'Gara P, Taubert KA; American Heart Association Committee on Rheumatic Fever, Endocarditis, and Kawasaki Disease of the Council on Cardiovascular Disease in the Young, Council on Clinical Cardiology, Council on Cardiovascular Surgery and Anesthesia, and Stroke Council. Infective Endocarditis in Adults: Diagnosis, Antimicrobial Therapy, and Management of Complications: A Scientific Statement for Healthcare Professionals From the American Heart Association. Circulation. 2015 Oct 13;132(15):1435-86. doi: 10.1161/CIR.0000000000000296. Epub 2015 Sep 15. PMID 26373316
- [Background] Pant S, Patel NJ, Deshmukh A, Golwala H, Patel N, Badheka A, Hirsch GA, Mehta JL. Trends in infective endocarditis incidence, microbiology, and valve replacement in the United States from 2000 to 2011. J Am Coll Cardiol. 2015 May 19;65(19):2070-6. doi: 10.1016/j.jacc.2015.03.518. PMID 25975469
- [Background] Habib G, Lancellotti P, Erba PA, Sadeghpour A, Meshaal M, Sambola A, Furnaz S, Citro R, Ternacle J, Donal E, Cosyns B, Popescu B, Iung B, Prendergast B, Laroche C, Tornos P, Pazdernik M, Maggioni A, Gale CP; EURO-ENDO Investigators. The ESC-EORP EURO-ENDO (European Infective Endocarditis) registry. Eur Heart J Qual Care Clin Outcomes. 2019 Jul 1;5(3):202-207. doi: 10.1093/ehjqcco/qcz018. PMID 30957862
- [Background] Habib G, Erba PA, Iung B, Donal E, Cosyns B, Laroche C, Popescu BA, Prendergast B, Tornos P, Sadeghpour A, Oliver L, Vaskelyte JJ, Sow R, Axler O, Maggioni AP, Lancellotti P; EURO-ENDO Investigators. Clinical presentation, aetiology and outcome of infective endocarditis. Results of the ESC-EORP EURO-ENDO (European infective endocarditis) registry: a prospective cohort study. Eur Heart J. 2019 Oct 14;40(39):3222-3232. doi: 10.1093/eurheartj/ehz620. PMID 31504413
- [Background] Dickerman SA, Abrutyn E, Barsic B, Bouza E, Cecchi E, Moreno A, Doco-Lecompte T, Eisen DP, Fortes CQ, Fowler VG Jr, Lerakis S, Miro JM, Pappas P, Peterson GE, Rubinstein E, Sexton DJ, Suter F, Tornos P, Verhagen DW, Cabell CH; ICE Investigators. The relationship between the initiation of antimicrobial therapy and the incidence of stroke in infective endocarditis: an analysis from the ICE Prospective Cohort Study (ICE-PCS). Am Heart J. 2007 Dec;154(6):1086-94. doi: 10.1016/j.ahj.2007.07.023. Epub 2007 Sep 12. PMID 18035080
- [Background] Nihoyannopoulos P, Oakley CM, Exadactylos N, Ribeiro P, Westaby S, Foale RA. Duration of symptoms and the effects of a more aggressive surgical policy: two factors affecting prognosis of infective endocarditis. Eur Heart J. 1985 May;6(5):380-90. doi: 10.1093/oxfordjournals.eurheartj.a061876. PMID 4043095
- [Background] Lodise TP, McKinnon PS, Swiderski L, Rybak MJ. Outcomes analysis of delayed antibiotic treatment for hospital-acquired Staphylococcus aureus bacteremia. Clin Infect Dis. 2003 Jun 1;36(11):1418-23. doi: 10.1086/375057. Epub 2003 May 20. PMID 12766837
- [Background] Shrestha NK, Ledtke CS, Wang H, Fraser TG, Rehm SJ, Hussain ST, Pettersson GB, Blackstone EH, Gordon SM. Heart valve culture and sequencing to identify the infective endocarditis pathogen in surgically treated patients. Ann Thorac Surg. 2015 Jan;99(1):33-7. doi: 10.1016/j.athoracsur.2014.07.028. Epub 2014 Oct 22. PMID 25442997
- [Background] Morris AJ, Drinkovic D, Pottumarthy S, Strickett MG, MacCulloch D, Lambie N, Kerr AR. Gram stain, culture, and histopathological examination findings for heart valves removed because of infective endocarditis. Clin Infect Dis. 2003 Mar 15;36(6):697-704. doi: 10.1086/367842. Epub 2003 Mar 4. PMID 12627353
- [Background] Lamas CC, Fournier PE, Zappa M, Brandao TJ, Januario-da-Silva CA, Correia MG, Barbosa GI, Golebiovski WF, Weksler C, Lepidi H, Raoult D. Diagnosis of blood culture-negative endocarditis and clinical comparison between blood culture-negative and blood culture-positive cases. Infection. 2016 Aug;44(4):459-66. doi: 10.1007/s15010-015-0863-x. Epub 2015 Dec 15. PMID 26670038
- [Background] Zegri-Reiriz I, de Alarcon A, Munoz P, Martinez Selles M, Gonzalez-Ramallo V, Miro JM, Falces C, Gonzalez Rico C, Kortajarena Urkola X, Lepe JA, Rodriguez Alvarez R, Reguera Iglesias JM, Navas E, Dominguez F, Garcia-Pavia P; Spanish Collaboration on Endocarditis-Grupo de Apoyo al Manejo de la Endocarditis infecciosa en Espana (GAMES). Infective Endocarditis in Patients With Bicuspid Aortic Valve or Mitral Valve Prolapse. J Am Coll Cardiol. 2018 Jun 19;71(24):2731-2740. doi: 10.1016/j.jacc.2018.03.534. PMID 29903346
- [Background] Fontana C, Favaro M, Pelliccioni M, Pistoia ES, Favalli C. Use of the MicroSeq 500 16S rRNA gene-based sequencing for identification of bacterial isolates that commercial automated systems failed to identify correctly. J Clin Microbiol. 2005 Feb;43(2):615-9. doi: 10.1128/JCM.43.2.615-619.2005. PMID 15695654
- [Background] Mignard S, Flandrois JP. 16S rRNA sequencing in routine bacterial identification: a 30-month experiment. J Microbiol Methods. 2006 Dec;67(3):574-81. doi: 10.1016/j.mimet.2006.05.009. Epub 2006 Jul 21. PMID 16859787
- [Background] Akram A, Maley M, Gosbell I, Nguyen T, Chavada R. Utility of 16S rRNA PCR performed on clinical specimens in patient management. Int J Infect Dis. 2017 Apr;57:144-149. doi: 10.1016/j.ijid.2017.02.006. Epub 2017 Feb 16. PMID 28216180
- [Derived] Pavone N, Cammertoni F, Calabrese M, Bruno P, Scoppettuolo G, Lombardo A, Giovannenze F, Taddei E, Fiori B, D'Inzeo T, Cutrone G, Iannaccone G, Del Zanna N, Massetti M. The expanding role of 16s ribosomal RNA PCR in the management of patients with infective endocarditis undergoing cardiac surgery. Front Cardiovasc Med. 2024 Dec 18;11:1504197. doi: 10.3389/fcvm.2024.1504197. eCollection 2024. PMID 39744206